# Title: Addressing ACEs Among Hispanic Caregivers in a Pediatric Primary Care Population to Improve Child Health and Decrease Early Adversity

NCT#: NCT05013138

Date: 08/25/2021

## You Are Being Asked to Be in a Research Study

Concise presentation of key concepts

You are being asked to be in a research study. A research study is designed to answer a scientific question. If you agree to be in the study you will be one of 840 people who are being studied, at Emory.

## Why is this study being done?

This study is being done to answer the question: How do childhood experiences affect parenting? You are being asked to be in this research study because you are receiving care at Mercy Care Chamblee for your new baby.

## Do you have to be in the study?

It is your decision to be part of this research study. You do not have to be in it. Your choice will not affect your access to medical care for your condition. Before you make your decision, you should take time to learn about the study.

## What do I have to do if I choose to participate in this study?

If you are eligible and want to be part of the study, you will answer questions about yourself and your child today. We will also contact you about 1 week, 6 months, and 18 months after today for more questions. The researchers will ask you to answer some questions about yourself.

## How is this study going to help you?

If you are in the study, you will be helping the researchers answer the study question.

## What are the risks or discomforts I should know about before making a decision?

The study will take time. Some questions may make you feel uncomfortable. All studies have some risks. Some risks are relatively small, like being bored or losing time. Some are more serious – for this study, these include distress when thinking about things that can be upsetting, loss of privacy, and breach of confidentiality. A full list of expected risks, their frequency and severity are in the "What are the possible risks and discomforts?" section of this document.

## Alternatives to Joining This Study

If you decide not to enter this study, you will still receive care by the Mercy Care Clinic and there is no effect to your treatment there by participating in this study.

Version Date: 07/10/2020



#### **Costs**

You WILL NOT have to pay for any of the study procedures.

### What Should I Do Next?

Read this form, or have it read to you. Make sure the study staff explains the study to you. Ask questions (e.g., about exact time commitment, about unfamiliar words, more details on specific procedures, etc.). Take time to consider this, and talk about it with your family and friends.




## Emory University Consent to be a Research Subject / HIPAA Authorization

<u>Title</u>: Addressing ACEs among Hispanic Caregivers in a Pediatric Primary Care Population to Improve Child Health and Decrease Early Adversity

IRB #: STUDY00002897

**Principal Investigator:** Abigail Powers Lott, PhD, ABPP

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### What is the purpose of this study?

The purpose of this study is to test whether being screened for adverse childhood experiences and having a conversation with your provider about your scores will improve health outcomes for your child versus just being screened for adverse childhood experiences.

#### What will I be asked to do?

If you agree to participate in the study, you will complete a series of questionnaires that ask about past adverse experiences, resilience, parenting, and psychological symptoms. This will take about 15-20 minutes. You will then either have a conversation with your provider about the information you provided or you will just have a usual wellness check visit for your child. Then, you will be contacted for follow up assessments that ask about resilience, parenting, and psychological symptoms 1 week, 6 months, and 18 months after your first visit. Each of these encounters will take about 15-20 minutes to complete. We will also look at the medical records of your infant to see how many medical visits they have during the course of the study.


 IRB Form 06162020



#### Who owns my study information and samples?

If you join this study, you will be donating your samples and study information. You will not receive any compensation if your samples or information are used to make a new product. If you withdraw from the study, data and samples that were already collected may be still be used for this study.

#### What are the possible risks and discomforts?

The most common risks and discomforts expected in this study are:

- -The risk of a loss of confidentiality
- -The risk of psychological distress when answering questions and discussing difficult experiences.

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

#### Will I benefit directly from the study?

This study is not designed to benefit you directly. This study is designed to learn more about if screening for adverse childhood experiences and provider-led discussions about those experiences help to improve child health outcomes. The study results may be used to help others in the future.

#### Will I be compensated for my time and effort?

All participants will have the ability to enter into our giveaways. You will get a giveaway entry for each component of the study you finish, with a total of up to 4 entries. If you decide to drop out of the study prior to getting a giveaway entry, you may still be entered into the giveaway by emailing Dr. Abigail Lott at adpower@emory.edu and Dr. Lott will add your entry into the giveaway. Twice during the course of the study, the study team will draw winning giveaway tickets for gift cards ranging from \$5-\$20. You will be alerted if you have one of the winning giveaway entries and will be given your prize. See Giveaway Official Rules for full details.

#### What are my other options?

If you decide not to enter this study, nothing will change about your pediatric primary care visit and we can still provide you with a resource packet of helpful resources.

#### How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

#### **Certificate of Confidentiality**

There is a Certificate of Confidentiality from the Center for Disease Control for this Study. The Certificate of Confidentiality helps us to keep others from learning that you participated in this study. Emory will rely on the Certificate of Confidentiality to refuse to give out study information that identifies you. For example, if Emory received a subpoena for study records, it would not give out information that identifies you.

The Certificate of Confidentiality does not stop you or someone else, like a member of your family, from giving out information about your participation in this study. For example, if you let your insurance company know that you are in this study, and you agree to give the insurance company research information, then the investigator cannot use the Certificate to withhold this information. This means you and your family also need to protect your own privacy.

The Certificate does not stop Emory from making the following disclosures about you:




- Giving state public health officials information about certain infectious diseases,
- Giving law officials information about abuse of a child, elderly person or disabled person.
- Giving out information to prevent harm to you or others.

Giving the study sponsor or funders information about the study, including information for an audit or evaluation.

#### **Storing and Sharing your Information**

De-identified data from this study (data that has been stripped of all information that can identify you), may be shared with the research community at large to advance science and health. Data from this study may be placed into public databases where, in addition to having no direct identifiers, researchers will need to sign data use agreements before accessing the data. We will remove or code any personal information that could identify you before your information is shared. This will ensure that, by current scientific standards and known methods, it is extremely unlikely that anyone would be able to identify you from the information we share. Despite these measures, we cannot guarantee anonymity of your personal data.

Your data from this study may be useful for other research being done by investigators at Emory or elsewhere. To help further science, we may provide your deidentified data to other researchers. If we do, we will not include any information that could identify you. If your data are labeled with your study ID, we will not allow the other investigators to link that ID to your identifiable information.

We will use your data only for research. We will not sell them. However, the results of this research might someday lead to the development of products (such as a specific therapy) that could be sold by a company. You will not receive money from the sale of any such product.

In general, we will not give you any individual results from the study of data you give us. If we find something of urgent medical importance to you, we will inform you, although we do not expect this to happen.

#### In Case of Injury

If you get ill or injured from being in the study, Emory will help you get treatment. Emory and the sponsor have not, however, set aside any money to pay you or to pay for this medical treatment. The only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory or sponsor employee. "Negligence" is the failure to follow a standard duty of care.

If you become ill or injured from being in this study, your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurer does not pay, then you will have to pay these costs.

If you believe you have become ill or injured from this research, you should contact Dr. Lott at telephone number



#### **Costs**

There will be no costs to you for participating in this study. You will not be charged for any of the research activities.

#### Withdrawal from the Study

You have the right to leave a study at any time without penalty.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.




#### Authorization to Use and Disclose Protected Health Information

The privacy of your health information is important to us. As part of this study, we will be requesting health care entities who are covered by the Health Insurance Portability and Accountability Act and regulations (HIPAA) to provide us with health information that identifies you ("individually identifiable health information" or "IIHI"). Because the health care entities are covered by HIPAA, we must have your authorization to obtain your IIHI from them. However, the researchers who get your IIHI from the health care entities are not covered by HIPAA. Once they receive your IIHI from the health care entities, they will put it in a separate research record that is not a part of your medical record. IIHI placed in the separate research record is not be covered by HIPAA.

#### **Purpose of this Authorization:**

By signing this form, you give us permission to get your IIHI from health care entities and to use and share your IIHI as described in this document. You do not have to sign this form. If you do not sign this form, then you may not participate in the research study.

#### **Research-Related Treatment**

This study involved research-related treatment that will not be electronically billed to any insurance company or government benefits program (e.g., Medicare, Medicaid). You may not receive the research-related treatment unless you sign this authorization. You may receive any non-research related treatment whether or not you sign this form.

#### IIHI that Will be Used/Disclosed:

The IIHI that we will use or share for the research study includes:

- Medical information about your infant including your infant's medical history and present/past medications.
- Number of infant's medical visits attended and the reason for those medical visits.

#### Purposes for Which Your IIHI Will be Used/Disclosed:

We will use and share your IIHI for the conduct and oversight of the research study. Once we have your IIHI we will keep it in a separate research record that will be used for the conduct of the study. If you leave the study, we may use your IIHI to determine your vital status or contact information.

#### Use and Disclosure of Your IIHI That is Required by Law:

We will use and disclose your IIHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults.

#### People Who will Use/Disclose Your IIHI:

The following people and groups will use and disclose your IIHI in connection with the research study:

- The Principal Investigator and the research staff will use and disclose your IIHI to conduct the study.
- The Principal Investigator and research staff will share your IIHI with other people and groups to help conduct the study or to provide oversight for the study. This includes sharing your IIHI with people and groups at other sites who are helping conduct the study.
- The Center for Disease Control and Prevention is the Sponsor of the study. The Sponsor may use and disclose your IIHI to make sure the research is done correctly and to collect and analyze the results of




the research. The Sponsor may disclose your IIHI to other people and groups like study monitors to help conduct the study or to provide oversight for the study.

- The following people and groups will use your IIHI to make sure the research is done correctly and safely:
  - Emory offices that are part of the Human Research Participant Protection Program and those that are involved in study administration. These include the Emory IRB, the Emory University and Healthcare Compliance Offices, and the Emory Office for Clinical Research.
  - Government agencies that regulate the research including: Office for Human Research Protections.
  - Research monitors and reviewer.
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your IIHI may be shared with that new institution and their oversight offices.

#### **Expiration of Your Authorization**

Your IIHI will be used until this research study ends.

#### **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your IIHI. If you want to do this, you must contact the study team at: Abigail Lott, 49 Jesse Hill Jr. Drive SE, Atlanta, GA 30303

At that point, the researchers would not collect any more of your IIHI. But they may use or disclose the information you already gave them as described in this Authorization. If you revoke your authorization you will not be able to stay in the study.

#### Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. HIPAA does not apply to research that does not include treatment that is billed to insurers or government benefit programs. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them. The researchers and people and companies working with them are not covered by the Privacy Rules. They will only use and disclose your information as described in this Consent and Authorization.

To maintain the integrity of this research study, you generally will not have access to your IIHI related to this research until the study is complete. When the study ends, and at your request, you generally will only have access to your IIHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. You will not have a right of access to IIHI kept in a separate research record used only for research purposed. If it is necessary for your health care, your health information will be provided to your doctor.

We may remove identifying information from your IIHI. Information without identifiers is not subject to HIPAA and may be used or disclosed with other people or organizations for purposes besides this study.

#### **Contact Information**

Contact Abigail Lott, PhD, ABPP at

- if you have any questions about this study or your part in it OR
- if you have questions, or concerns about the research

Contact the Emory Institutional Review Board at




- if you have questions about your rights as a research participant.
- if you have complaints about the research or an issue you rather discuss with someone outside the research team.

You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="https://tinyurl.com/ycewgkke">https://tinyurl.com/ycewgkke</a>.




## **Consent and Authorization**

| TO BE FILLED OUT BY SUBJECT ONLY | | | |
|---|---|---|---|
| Please <b>print</b> your name, <b>sign</b> , and <b>date</b> below if you agree to be in the stu | | consent and author | ization |
| form, you will not give up any of your legal rights. We will give you a copy of | the form to keep. | | |
| Name of Infant | - | | |
| | - | | |
| Name of Subject | | | |
| Signature of Subject (18 or older and able to consent) | Date | Time | |
| TO BE FILLED OUT BY STUDY TEAI | M ONLY | | |
| Name of Person Conducting Informed Consent Discussion | | | |
| Signature of Person Conducting Informed Consent Discussion | Date | Time | |
